CLINICAL TRIAL: NCT07201571
Title: A Retrospective Cohort Study of Patients Who Underwent Curative-intent Esophagectomy for ESCC at a Tertiary Referral Center in South Korea
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seong Yong Park, Samsung Medical Center, Samsung Medical Center
Other Study IDs: SMC-ESCC
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Oesophageal Squamous Cell Carcinoma
Keywords: Oesophageal Squamous Cell Carcinoma; Esophagectomy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent curative surgery for esophageal cancer: Patients who underwent curative surgery for esophageal cancer

SUMMARY:
This retrospective cohort study was conducted using the Registry for Thoracic Cancer Surgery at Samsung Medical Center (Seoul, South Korea), which has included all patients who underwent thoracic surgery

DETAILED DESCRIPTION:
This retrospective cohort study was conducted using the Registry for Thoracic Cancer Surgery at Samsung Medical Center (Seoul, South Korea), which has included all patients who underwent thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent curative surgery for esophageal cancer

Exclusion Criteria:

* cervical esophageal cancer
* gastroesophageal junction cancer
* histology other than squamous cell carcinoma
* patients with Child-Pugh class B or C liver cirrhosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent curative surgery for esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 3131 (Actual)
Dates: Start 1994-11-06 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | within 90 days after surgery
  Complications related to fluid imbalance and portal hypertension, such as ascites, pleural effusion, and chyle leak; complications associated with impaired renal or hematologic function, including acute kidney injury, bleeding, and graft failure; and complications reflecting immune dysfunction and infection susceptibility, including pneumonia and empyema. Complications associated with impaired tissue healing, such as anastomotic leakage, were also analyzed. Liver failure and acute respiratory distress syndrome were considered separately. All complications were defined according to the Esophageal Complications Consensus Group, and their severity was assessed according to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Overall survival | 10 years after surgery
  Interval from the date of surgery to death or censoring

IPD SHARING:
Plan to Share IPD: Undecided